CLINICAL TRIAL: NCT06373237
Title: Retrospective Observation of Outcomes of Embryos Transferred After Initial Chaotic Results on Preimplantation Genetic Testing for Aneuploidy (PGT-A)
Brief Title: Outcome of Embryos Transferred After Initial Chaotic Results on PGT-A
Status: Completed | Type: Observational
Sponsor: Inception Fertility Research Institute, LLC (Industry)
Collaborators: Igenomix (Industry)
Responsible Party: Sponsor
Other Study IDs: INC-IG-2024-001
Record Dates: First submitted 2024-04-08; First posted 2024-04-18 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a retrospective review of treatment outcomes from fertility clinics in The Prelude Network who have used Igenomix for PGT-A and have transferred embryos with initial chaotic results, regardless if re-biopsy was performed.

DETAILED DESCRIPTION:
Primary objective: to observe the outcomes of embryos transferred with initial "chaotic" results on PGT-A via Igenomix.

Hypothesis: The transfer of chaotic embryos can result in clinical pregnancy, as defined by fetal heartbeat at 6-8 weeks gestation. Furthermore, these transfers may also result in live birth and expand reproductive potential for patients seeking IVF with PGT-A.

ELIGIBILITY:
Inclusion Criteria:

* Patients that conducted PGT-A via Igenomix who have transferred an embryo with an initial chaotic result.

Exclusion Criteria:

* Patients who had multiple embryo transfer.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women of any age who have conducted PGT-A via Igenomix who have transferred an embryo with an initial chaotic result.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2024-03-26 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
Embryo re-biopsy rate | 2 years
  Frequency of re-biopsy post initial chaotic PGT-A result
Embryo transfer rate | 2 years
  Frequency of embryo transfer post re-biopsy
Pregnancy rate | 2 years
  Frequency of positive serum pregnancy test post embryo transfer of initial chaotic embryo
Live birth rate | 2 years
  Frequency of live birth post embryo transfer of initial chaotic embryo

CONTACTS AND LOCATIONS:
Locations (1):
- Inception Fertility LLC, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No